CLINICAL TRIAL: NCT00594269
Title: Discontinuation of Antipsychotics and Antidepressants Among Patients With Dementia and BPSD Living in Nursing Homes - a 24 Weeks Double Blind RCT.
Brief Title: Dementia Antipsychotics And Antidepressants Discontinuation Study
Acronym: DESEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Ullevaal University Hospital (Other); Eikertun Nursing Home (Other); University of Bergen (Other); Innlandet Hospital Trust, Sanderud (Unknown); Innlandet Hospital Trust, Reinsvoll (Unknown); Diakonhjemmet Hospital (Other); Sykehuset Telemark (Other Government); The Nordmøre and Romsdal Hospital Trust (Unknown); Songdalstunet Nursing Home (Other); Sykehuset Buskerud HF (Other); Kroken Nursing Home, Tromsø (Other); Kløveråsen, Bodø (Unknown); Bjørgene Omsorgssenter, Haugesund (Unknown); Alesund Hospital (Other)
Responsible Party: Sverre Bergh, Cand Med, Researcher., Innlandet Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F06001
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Dementia
Keywords: Antidepressants; Antipsychotics; Dementia; Discontinuation study; Behavioural- and Psychological Symptoms in Dementia
MeSH Terms: conditions — Dementia | interventions — Risperidone; Escitalopram; Citalopram; Sertraline; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator): Discontinuation of antipsychotic or antidepressants
  Interventions: Drug: Risperidone; Drug: Escitalopram; Drug: Citalopram; Drug: Sertraline; Drug: Paroxetine

INTERVENTIONS:
Drug: Risperidone — Discontinuation
  Other Names: ATC code N05AX 08
Drug: Escitalopram — Discontinuation
  Other Names: ATC code N06AB 10
Drug: Citalopram — Discontinuation
  Other Names: ATC code N06AB 04
Drug: Sertraline — Discontinuation
  Other Names: ATC code N06AB 06
Drug: Paroxetine — Discontinuation
  Other Names: ATC code N06AB 05

SUMMARY:
The aim of this study is to discontinue antipsychotics and antidepressants, and to study its effect on Behavioural- and Psychological Symptoms in Dementia (BPSD).

DETAILED DESCRIPTION:
Patients with dementia have cognitive deficits, but also hallucinations, delusions, agitation, aggression and apathy. These symptoms are called Behavioural- and Psychological Symptoms in Dementia (BPSD), and are difficult to treat. Antipsychotic and antidepressant medication is used as treatment, despite its lack of clinical evidence.

We will discontinue risperidone in one group of 30 patients and compere them to 30 controls and we will discontinue antidepressants in a group of 76 patients and compere them to 76 controls. Patients should have dementia of Alzheimer- or vascular origin. They should live in Nursing Homes and have no other psychiatric disease for which they receive psychotropic drug. They will be registered with 7 different questionnaires at baseline and after 3, 6, 12 and 24 weeks. The study period is 24 weeks. The questionnaires are filled in by the patients and the nurses at the nursing homes.

This is a double blind RCT study with placebo-controlled group.

ELIGIBILITY:
Inclusion Criteria:

* Vascular- or Alzheimer Dementia
* Nursing Homes resident for 3 months or more
* Given antipsychotics or antidepressants for 3 months or more
* Clinical Dementia rating 1, 2 or 3

Exclusion Criteria:

* Dementia of other origin
* Psychiatric disease
* Life expectancy less than 3 months
* Acute infection last 10 days
* Unstable Diabetes Mellitus
* Terminal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in Neuropsychiatric Inventory | 24 weeks
Changes in Cornell's Depression Scale | 24 weeks
Changes in UPDRS subscale | 24 weeks

SECONDARY OUTCOMES:
Changes in Severe Impairment Battery | 24 weeks
Changes in Lawton's PADL | 24 weeks
Oxazepam given p.n. | 24 weeks
Number of falls | 24 weeks
Changes in Body Weight | 24 weeks
Quality of Life - Alzheimer disease | 24 weeks
Clinical Dementia Rating | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, Ph D, Study Chair — The Norwegian Centre for Dementia Research (NCDR), Norway; Sverre Bergh, MD, Principal Investigator — Innlandet Hospital Trust, Sanderud
Locations (8):
- Norway (8):
  - Sykehuset Innlandet HF - Sanderud, Ottestad, Oppland
  - Sykehuset Innlandet HF, Reinsvoll, Oppland
  - University of Bergen, Løvaasen Nursing Home, Bergen
  - Eikertun Nursing Home, Hokksund
  - The Nordmøre and Romsdal Hospital Trust, Molde
  - Diakonihjemmets Hospital, Oslo
  - Ullevaal University Hospital, Oslo
  - Telemark Hospital, Skien

REFERENCES:
- [Derived] Bergh S, Selbaek G, Engedal K. Discontinuation of antidepressants in people with dementia and neuropsychiatric symptoms (DESEP study): double blind, randomised, parallel group, placebo controlled trial. BMJ. 2012 Mar 9;344:e1566. doi: 10.1136/bmj.e1566. PMID 22408266